CLINICAL TRIAL: NCT01919489
Title: A Randomized Controlled Trial Comparing the Safety and Efficacy of Liraglutide Versus Glargine Insulin for the Management of Patients With Type 2 Diabetes After Hospital Discharge
Brief Title: Liraglutide Hospital Discharge Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Novo Nordisk A/S (Industry)
Responsible Party: Principal Investigator, Guillermo Umpierrez, MD, Professor of Medicine, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00068128; (UTN) U1111-1139-2991 (Registry Identifier: UNIVERSAL TRIAL NUMBER)
Record Dates: First submitted 2013-07-30; First posted 2013-08-09 (Estimated); Results first posted 2021-11-03 (Actual); Last update posted 2021-11-03 (Actual); Status verified 2021-08

CONDITIONS: Type 2 Diabetes
Keywords: Incretins; Liraglutide; Glargine; Randomized controlled trial; basal insulin; hospital discharge; inpatient diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Liraglutide; Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Liraglutide + OADs (Experimental): Liraglutide once daily in combination to oral anti-diabetic agents (OADs)
  Interventions: Drug: Liraglutide + OADs
- Glargine + OADs (Active Comparator): Glargine once daily in combination to oral anti-diabetic agents (OADs)
  Interventions: Drug: Glargine + OADs

INTERVENTIONS:
Drug: Liraglutide + OADs — Liraglutide subcutaneously daily
  Other Names: Victoza® + OADs
  Arms: Liraglutide + OADs
Drug: Glargine + OADs — Glargine once daily subcutaneously
  Other Names: Glargine (Lantus®) + OADs
  Arms: Glargine + OADs

SUMMARY:
High blood glucose levels in hospitalized patients with diabetes are associated with increased risk of medical complications and death. Improved glucose control with insulin injections may improve clinical outcome and prevent some of the hospital complications. Increasing evidence indicates that incretin-based agents are safe and effective for the hospital management of patients with type 2 diabetes (T2D).

Liraglutide is a once-daily human glucagon-like peptide (GLP-1) analogue approved for the treatment of T2D. Liraglutide has been shown to lower blood glucose, stimulate endogenous insulin secretion, decrease plasma glucagon levels, inhibit gastric emptying, reduce food intake and body weight and improve ß-cell function when administered subcutaneously. Liraglutide increases insulin secretion in a glucose-dependent manner (i.e., only when plasma glucose levels are elevated), resulting in low-risk of hypoglycemia when used as monotherapy. When compared to insulin glargine therapy, the use of GLP-1 has resulted in comparable reduction in HbA1c level, lower rates of hypoglycemia and less weight gain. No prospective studies; however, have compared the efficacy and safety of liraglutide in the hospital setting or after hospital discharge.

The primary objective is to compare the safety and efficacy of liraglutide (Victoza®) versus glargine insulin in combination to oral anti-diabetic agents (OADs: metformin, sulfonylureas, nateglinide, repaglinide or pioglitazone) on glycemic control after 26 weeks of treatment in medicine patients with T2D after hospital discharge.

DETAILED DESCRIPTION:
Specific Aim: To determine whether treatment with liraglutide (Victoza®) will result in similar glycemic control (HbA1c at 26 weeks) and a lower rate of hypoglycemic events compared to treatment with glargine (Lantus®) in patients with T2D after hospital discharge. Patients with poorly controlled (HbA1c >7%-10%) T2D treated with diet or oral antidiabetic agents or low dose insulin naïve (0.4u/kg/day) prior to admission will be randomized to liraglutide or glargine in combination to OADs at hospital discharge.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females between the ages of 18 and 80 years discharged after hospital admission from non- ICU general surgery and medicine services (excluding gastrointestinal and cardiac surgeries).
2. Admission HbA1c between 7% and 10%
3. Patients with T2D treated with diet alone or with oral antidiabetic agents as monotherapy or in combination therapy (excluding GLP1 receptor agonists) or on low-dose insulin therapy (TDD ≤0.4 unit/kg/day) prior to admission.
4. Subjects with a hospital admission BG < 400 mg/dL without laboratory evidence of diabetic ketoacidosis (serum bicarbonate < 18 mEq/L or positive serum or urinary ketones).
5. BMI > 25 Kg/m2 and ≤ 45 Kg/m2

Exclusion Criteria:

1. Age < 18 or > 80 years.
2. Subjects with stress hyperglycemia (BG > 140 mg/dL and HbA1c < 6.5%)
3. Subjects with a history of type 1 diabetes
4. Treatment with insulin or GLP-1 analogs during the past 3 months prior to admission.
5. Recurrent severe hypoglycemia or hypoglycemic unawareness.
6. Subjects with gastrointestinal obstruction, gastroparesis, or those expected to require gastrointestinal suction.
7. History of medullary thyroid cancer or multiple endocrine neoplasias
8. Patients with acute or chronic pancreatitis, pancreatic cancer, or gallbladder disease.
9. Patients with clinically significant hepatic disease (cirrhosis, jaundice, end-stage liver disease, portal hypertension) and elevated ALT and AST > 3 times upper limit of normal, or significantly impaired renal function (GFR < 30 ml/min).
10. Treatment with oral or injectable corticosteroid (equivalent or higher than prednisone 5mg/day), parenteral nutrition, and immunosuppressive treatment.
11. Mental condition rendering the subject unable to understand the nature, scope, and possible consequences of the study.
12. Female subjects who are pregnant or breastfeeding at the time of enrollment into the study.
13. Females of childbearing potential who are not using adequate contraceptive methods (as required by local law or practice).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 273 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2020-08-30 (Actual); Study Completion 2020-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo E Umpierrez, MD, Principal Investigator — Emory University SOM
Locations (5):
- United States (5):
  - University of Miami, Miami, Florida
  - Grady Memorial Hospital, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia
  - Emory Universtiy Hospital at MIdtown, Atlanta, Georgia
  - State University of NY at Buffalo, New York, New York

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Liraglutide + OADs | Glargine + OADs
Started | 136 | 137
Completed | 80 | 93
Not Completed | 56 | 44
Not completed — Rejected the need of injections | 4 | 7
Not completed — Adverse Event | 10 | 0
Not completed — Hospital readmission | 2 | 9
Not completed — Death | 2 | 1
Not completed — Lost to Follow-up | 38 | 27

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Liraglutide + OADs | Glargine + OADs | Total
Number analyzed (Participants) | 136 | 137 | 273
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.1 (9.5) | 55.9 (11.2) | 56.1 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 61 | 108
  Male | 89 | 76 | 165
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 97 | 95 | 192
  White | 23 | 27 | 50
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 16 | 15 | 31
Region of Enrollment [Number; unit: participants]
  United States | 133 | 134 | 267
  Argentina | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Glycemic Control at Hospital Discharge and 6 Months Follow up
Description: To determine differences in HbA1c concentration at 26 weeks from discharge between liraglutide and glargine insulin therapy
Time Frame: Hospital discharge, 6 months (26 weeks)
Population: Number of subjects analyzed at 6 months differs from overall number of subjects analyzed, due to patients unable to complete the trial: 56 in the Liraglutide Arm and 44 in the Glargine Arm.
Measure: Mean (Standard Deviation); unit: % (mmol/mol)
Arm/Group | Liraglutide + OADs | Glargine + OADs
Number analyzed (Participants) | 136 | 137
% (mmol/mol)
  HbA1C at hospital discharge | 8.3 (0.9) | 8.4 (0.8)
  HbA1C at 6 months post-intervention: number analyzed (Participants) | 80 | 93
  HbA1C at 6 months post-intervention | 7.13 (1.3) | 7.68 (1.69)

2. Secondary Outcome: Fasting and Postprandial Blood Glucose (BG) Concentration After Follow up of 26 Weeks
Description: To determine differences in BG concentration between liraglutide and glargine insulin therapy
Time Frame: After discharge, average at 3 months (12 week) and 6 months (26 weeks)
Population: The number of subjects analyzed in this outcome at different time points from the overall number of subjects analyzed in other timepoints because it includes only those participants who were able to provide blood glucose results at the specified time points reported (12 and 26 weeks).
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Liraglutide + OADs | Glargine + OADs
Number analyzed (Participants) | 60 | 79
mmol/L
  Fasting blood glucose at 26 weeks follow up | 7.61 (2.2) | 8.56 (3.8)
  Post-prandial blood glucose at 12 weeks: number analyzed (Participants) | 44 | 42
  Post-prandial blood glucose at 12 weeks | 7.67 (1.6) | 9.32 (8.8)
  Postprandial blood glucose at 26 weeks follow up: number analyzed (Participants) | 53 | 60
  Postprandial blood glucose at 26 weeks follow up | 8.23 (2.8) | 8.72 (2.3)
  Fasting blood glucose at 12 weeks | 7.96 (3.3) | 7.70 (2.6)

3. Secondary Outcome: Hypoglycemic Episodes
Description: Number of participants who had at least one hypoglycemic event (<70 mg/dl) and severe hypoglycemic event (<40 mg/dl)
Time Frame: After discharge, average 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Liraglutide + OADs | Glargine + OADs
Number analyzed (Participants) | 136 | 137
Participants
  Participants who had at least one hypoglycemic events (<70 mg/dl) | 18 | 31
  Participants who had at least one severe hypoglycemic event (<40 mg/dl) | 2 | 3

4. Secondary Outcome: HbA1c <7.0% and no Hypoglycemia
Description: Percent of patients with 26 week HbA1c <7.0% and no hypoglycemia
Time Frame: After discharge, average 6 months
Population: This outcome included only participants with available data for both variables: HbA1c and hypoglycemia
Measure: Count of Participants; unit: Participants
Arm/Group | Liraglutide + OADs | Glargine + OADs
Number analyzed (Participants) | 76 | 88
Participants | 34 | 29

5. Secondary Outcome: HbA1c <7.0% and no Weight Gain
Description: Percent of patients with 26 week HbA1c <7.0% and no weight gain
Time Frame: After discharge, average 6 months
Population: This outcome included only participants with available data for both variables: HbA1c and weight
Measure: Count of Participants; unit: Participants
Arm/Group | Liraglutide + OADs | Glargine + OADs
Number analyzed (Participants) | 78 | 90
Participants | 32 | 21

6. Secondary Outcome: HbA1c <7.0% and no Hypoglycemia
Description: Percent of patients with 12 week HbA1c <7.0% and no hypoglycemia
Time Frame: After discharge, average 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Liraglutide + OADs | Glargine + OADs
Number analyzed (Participants) | 83 | 94
Participants | 40 | 31

7. Secondary Outcome: Change in Body Weight From Baseline
Description: Change in body weight from baseline after 6 months of follow up (26 weeks)
Time Frame: After discharge, average 6 months
Population: This outcome only included participants with available data for body weight in Kgs at baseline and 26 weeks follow up.
Measure: Mean (Standard Deviation); unit: Kgs
Arm/Group | Liraglutide + OADs | Glargine + OADs
Number analyzed (Participants) | 73 | 91
Kgs
  Baseline weight at discharge | 101.0 (20.6) | 98.2 (18.0)
  Weight at six months | 97.2 (19.9) | 98.3 (22.1)
  Weight change from baseline (discharge) to 6 months after discharge | -4.77 (8) | 0.6 (11)

8. Secondary Outcome: Change in BMI
Description: Change in BMI after 6 months from baseline
Time Frame: Baseline, and follow up after discharge (average 6 months)
Population: This outcome only included participants with available data for BMI at baseline and follow up of 26 weeks.
Measure: Mean (Standard Deviation); unit: kg/m2
Arm/Group | Liraglutide + OADs | Glargine + OADs
Number analyzed (Participants) | 136 | 137
kg/m2
  Baseline BMI | 33.5 (5.3) | 33.3 (5.3)
  BMI at 26 weeks follow up: number analyzed (Participants) | 73 | 91
  BMI at 26 weeks follow up | 32.7 (6.8) | 33.3 (6.2)

9. Secondary Outcome: Total Daily Dose of Insulin
Description: Evaluate the total daily dose of insulin needed in the group receiving glargine
Time Frame: After discharge, average 6 months
Population: This outcome analyzed participants with available medication dose for the 26 weeks follow up.
Measure: Mean (Standard Deviation); unit: IU per day
Arm/Group | Liraglutide + OADs | Glargine + OADs
Number analyzed (Participants) | 73 | 90
IU per day | 0 (0) | 20.9 (11.1)

10. Secondary Outcome: Change in Cardiovascular Risk Factors: Blood Pressure
Description: Cardiovascular risk factors including changes in systolic and diastolic blood pressure from baseline to 26 weeks post-intervention
Time Frame: Baseline, 26 weeks post-intervention
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Liraglutide + OADs | Glargine + OADs
Number analyzed (Participants) | 73 | 90
mmHg
  Systolic blood pressure at baseline | 134 (17) | 130 (17)
  Systolic blood pressure at 26 weeks follow up | 136 (22) | 135 (19)
  Diastolic blood pressure at baseline | 79 (11) | 77 (12)
  Diastolic blood pressure at 26 weeks follow up | 80 (13) | 79 (14)

11. Secondary Outcome: Cardiovascular Risk Factor: Heart Rate
Description: Cardiovascular risk: heart rate at baseline and 26 weeks post-intervention
Time Frame: 26 weeks post-intervention
Population: This outcome included patients with available heart rate data at 26 weeks follow-up.
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | Liraglutide + OADs | Glargine + OADs
Number analyzed (Participants) | 73 | 90
beats/min
  Heart rate at baseline (discharge) | 79 (14) | 79 (14)
  Heart rate at 6 months post-discharge | 83 (13) | 79 (14)

12. Secondary Outcome: Cardiovascular Risk Factor: Lipid Profile
Description: Lipid profile was measured with total cholesterol level results at 26 weeks post-intervention. This outcome was not part of standard of care.
Time Frame: 26 weeks post-intervention
Population: Total cholesterol was measured in 9 subjects only due to limited funding.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Liraglutide + OADs | Glargine + OADs
Number analyzed (Participants) | 4 | 5
mg/dL | 190 (6) | 130 (56)

13. Secondary Outcome: Emergency Room Visits and Readmissions
Description: Number of participants who had at least one emergency room visit and hospital readmissions
Time Frame: After discharge, average 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Liraglutide + OADs | Glargine + OADs
Number analyzed (Participants) | 136 | 137
Participants
  Number of participants with at least one ER visit | 31 | 23
  Number of participants with at least one hospital readmission | 35 | 43

14. Secondary Outcome: Acute Renal Failure
Description: Acute renal failure during the 26-week follow-up defined as a clinical diagnosis of acute renal failure with documented new-onset abnormal renal function (increment in creatinine > 0.5 mg/dL from baseline)
Time Frame: After discharge, average 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Liraglutide + OADs | Glargine + OADs
Number analyzed (Participants) | 136 | 137
Participants | 1 | 3

15. Secondary Outcome: Self-measured Blood Glucose (SMBG) 7-point Profiles at 26 Weeks Follow up
Description: Number of participants that reported self-measured blood glucose (SMBG) 7-point profiles at 26 weeks follow up
Time Frame: 26 weeks post-intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Liraglutide + OADs | Glargine + OADs
Number analyzed (Participants) | 136 | 137
Participants | 34 | 34

ADVERSE EVENTS:
Time Frame: Data collected during follow up (6 months post-intervention).
Arm/Group | Liraglutide + OADs | Glargine + OADs
All-Cause Mortality (participants affected / at risk) | 2/136 | 1/137
Serious Adverse Events (participants affected / at risk) | 52/136 | 54/137
Other Adverse Events (participants affected / at risk) | 0/136 | 0/137
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Liraglutide + OADs (N=136) | Glargine + OADs (N=137)
Readmissions (General disorders) | 35 (60) | 43 (94)
Congestive heart failure (Cardiac disorders) | 12 (21) | 13 (34)
Medication discontinued due to AEs (General disorders) | 13 (13) | 0 (0)
Cerebrovascular event (Nervous system disorders) | 0 (0) | 3 (3)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 3 (3)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 37 (37) | 3 (3)
Vomiting (Gastrointestinal disorders) | 18 (18) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-28): https://cdn.clinicaltrials.gov/large-docs/89/NCT01919489/Prot_SAP_000.pdf